CLINICAL TRIAL: NCT05891301
Title: Construction and Validation of Risk Prediction Model for Gastrointestinal Dysfunction of Patient With Colorectal Cancer After Surgery
Brief Title: Construction and Validation of Risk Prediction Model for Gastrointestinal Dysfunction of Patient With Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Other Study IDs: cwd-M1
Record Dates: First submitted 2023-05-27; First posted 2023-06-06 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Patient With Colorectal Cancer; Surgery
Keywords: colorectal cancer; surgery; gastrointestinal dysfunction; risk prediction model
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- questionnaires assessed patient with colorectal cancer after surgery: Patients with colorectal cancer who had a radical resection surgery.
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — The contents of the questionnaire included gender, age, BMI, previous operation history, previous medication history, smoking history,patient mobility in the hospital, etc.Questionnaire was completed on the first postoperative day.From the third day to the end of the seventh day, patients were evaluated daily for gastrointestinal dysfunction.Postoperative mobility was assessed daily.

SUMMARY:
To understand the current situation of the postoperative gastrointestinal dysfunction in patients with colorectal cancer effect a radical cure, and analyze the risk factors, and build the colorectal cancer radical surgery in patients with gastrointestinal dysfunction risk prediction nomogram model decision tree classification and regression tree model, through internal validation evaluation the performance of the two models in the modeling data set and dividing the postoperative gastrointestinal dysfunction risk level.Two risk prediction models were used to carry out external verification, evaluate the clinical practicability and effectiveness of the model, and provide reference for further promotion of the model.

DETAILED DESCRIPTION:
Colorectal cancer is characterized by high morbidity and mortality. Surgical treatment is the main treatment for colorectal cancer. Surgery is the best treatment for long-term survival.

Surgery is a destructive operation, can lead to local tissue injury, physical barrier damage, causes the patient's body, and a series of metabolism, neuroendocrine and immune response, all of which can cause local inflammation or systemic inflammatory response, also leads to occurrence of related complications, such as abdominal and pelvic infection, fever, anastomotic infection and fistula, intestinal obstruction, etc., Thus increasing the risk of postoperative complications. The trauma and irritation of gastrointestinal tract caused postoperative gastrointestinal dysfunction.

The procedure of surgery is accompanied by anesthesia, and the anesthesia mode of gastrointestinal surgery is mainly general anesthesia. Opioid analgesics are one of the most important components of general anesthesia. The most common side effects of opioid analgesics include postoperative intestinal obstruction, nausea and vomiting, chills and urinary retention. The use of anesthetic drugs further aggravated the postoperative gastrointestinal dysfunction.

At the same time, laparoscopic surgery must establish pneumoperitoneum pressure. In recent years, studies have suggested that pneumoperitoneum pressure can lead to changes in the body's internal environment, resulting in a series of pathophysiological changes such as tissue ischemia, intestinal edema, and release of inflammatory factors in the gastrointestinal tract, resulting in dysfunction of gastrointestinal function.

All the above reasons lead to gastrointestinal dysfunction as the highest complication after radical resection of colorectal cancer.A review of previous literature shows that there is no predictive assessment tool for gastrointestinal dysfunction in patients after radical resection of colorectal cancer.Therefore, it is necessary to construct a risk prediction model for patients after radical resection of colorectal cancer, and to verify the clinical practicability of the model through external verification.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years;
* patients with diagnosed colon or rectal cancer;
* Patients diagnosed as having undergone radical resection of colorectal cancer;
* Patients who can read and communicate in Chinese.

Exclusion Criteria:

* Patients with multiple cancers;
* Patients who are unable to communicate due to dementia, language disorders or postoperative mental disorder or hearing impairment.

withdrawl Criteria：

* Patients with postoperative mechanical obstruction;
* Patients requiring reoperation for any indication prior to the initiation of formal evaluation of POGD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 516 cases needed to be included in the modeling group and 221 cases needed to be included in the validation group
Sampling Method: Probability Sample
Enrollment: 737 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
gastrointestinal dysfunction | 3 days after surgery
  The gastrointestinal dysfunction will be assessed by 《Intake, Feeling nauseated, Emesis, Exam, and Duration of symptoms scoring system(I-FEED)》.The questionnaire consisted of 5 items.The scale contains five items, with the highest score of 3 and the lowest score of 0 for each item. Items include: tolerance to eating, presence of nausea, presence of vomiting, presence of bloating, duration of symptoms.A score of 6 or greater is a diagnosis of gastrointestinal dysfunction.

SECONDARY OUTCOMES:
BMI | Baseline
  Weight/(Height)²
Smoking history | Baseline
  Smoking history will be assessed by 《Patient General Data Collection Form》,described by "yes" or "not".If patient has smoking history, the form will record how many cigarettes are smoked per day.
Nutritional Risk | Baseline
  It will be assessed by《European Nutritional Risk Screening 2002(NRS 2002)》.If the score ≥3, it indicates high nutritional risk.The scale contains three items, namely, disease severity, nutritional status, and age. Among them, the highest score of disease severity and nutritional status was 3 and the lowest score was 0. Age ≥70 years is one point.
Previous medication history | Baseline
  Medications history will be assessed by 《Patient General Data Collection Form》,described by "History of use of chemotherapeutics" 、"History of use of opiates"、"History of use of antithrombotic drugs" or "not".
Previous operation history | Baseline
  Previous operation history will be assessed by 《Patient General Data Collection Form》,described by "History of non-abdominal surgery" 、"History of colectomy surgery"、"History of rectotomy surgery"、"History of other abdominal surgery" or "none".
Preoperative bowel preparation | one day before surgery
  It will be assessed by 《Bristol stool form scale》.Divided into 7 types, type 1 stool is granular, difficult to discharge. Type 2 is salami, which is hard. Type 3 is a strip with a cracked surface. Type 4 is strip, smooth surface, soft texture, easy to discharge. Type 5 stools are clumpy and soft in texture. Type 6 is a mushy loose stool. Type 7 is watery stool.
Patient Mobility in the hospital | one day after surgery
  Patient Mobility l will be assessed by 《Inter-rater reliability of the Johns Hopkins Highest Level of Mobility Scale (JH-HLM)》.The maximum score of the scale is 8 points, 1 to 3 points means that only bed activities can be carried out, 4-5 points means that bedside activities can be carried out, and 6-8 points means that under-bed activities can be carried out. The higher the score, the higher the level of activity.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, Phd, Principal Investigator — Sun Yat-sun Unversity
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No